CLINICAL TRIAL: NCT00259324
Title: Childhood Obesity Treatment Targeting Specific Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-R21-DK07491901
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2007-12

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental): Diet and Activity
  Interventions: Behavioral: Diet and Activity
- 2 (Experimental): Diet and Activity
  Interventions: Behavioral: Diet and Activity
- 3 (Placebo Comparator): Education
  Interventions: Behavioral: Diet and Activity

INTERVENTIONS:
Behavioral: Diet and Activity — Diet and Activity

SUMMARY:
The US is in the midst of an obesity epidemic, affecting young children. The pediatric primary care setting is an ideal place to address this problem since most families have frequent contact with their pediatrician and a child's health status is regularly assessed in this setting. Recommendations for treating children with a body mass index (BMI) over the 85th percentile in the primary care setting have been developed by an Expert Committee on childhood. Programs are needed that meet the recommendations from the Committee, which include: 1) beginning treatment as young as possible; 2) focusing on the family, with the parent being the primary change agent for treatment; 3) using behavior modification techniques to change eating and activity behaviors; and 4) making 2 or 3 very specific changes in diet and activity at one time. Thus, the aim of this R21 application is to develop, implement, and evaluate a 6-month behavioral childhood obesity intervention that meets the Committee's recommendations and can be implemented in a primary care setting. A second aim of this project is to determine which eating and activity behaviors should be targeted in the intervention. One hundred thirty-five children, aged 4 to 9 years with a BMI > 85th percentile, assessed and referred by their pediatricians, will be randomized to one of three conditions: 1) a newsletter condition; 2) a Behavioral Parenting Program that increases physical activity (60 min/day) and decreases sweetened drink consumption (< 3 servings/week) (Traditional); or 3) a Behavioral Parenting Program that reduces TV watching (< 2 hours/day) and increases low-fat milk consumption (2 servings/day) (Substitutes). Follow-up assessments on weight, height, and standardized BMI (z-BMI), the primary dependent variable, will be conducted at 3, 6, 9, and 12 months. Pediatricians will provide follow-up letters to families, regarding weight and height status, following the assessments. This pilot study allows us to determine the feasibility and efficacy of a pediatric obesity intervention that optimizes the role of the pediatrician and meets the Committee's recommendations for treatment in a primary care setting. Moreover, by comparing the effects of targeting the traditional or substitute behaviors, data will be obtained for a power analysis for a full-scale trial of the effects of these two approaches on long-term weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age between 4 and 9 years. We propose to use this age group since parents are in control of the eating and exercise choices of such children, and thus a program that focuses on parenting behaviors (i.e., positive reinforcement, stimulus control, parental modeling) should be developmentally appropriate. This age group also meets the Expert Committee's goal of intervening early5; moreover children aged 4 to 8 years have similar nutritional needs.

  2) Body mass index (BMI) > 85th percentile BMI. Based upon the Expert Committee recommendations,5 children > 2 years of age who are identified as being at risk for overweight (85th to 94th percentile BMI) or overweight (> 95th percentile BMI) should focus on weight maintenance as height continues to increase. These recommendations are aimed at reducing z-BMI.

  3) Tanner stage 1 (prepubertal) sexual maturation status. 4) Self-report at least one of the following problematic behaviors:
  1. Consume > 1 serving of sweetened drink per day.
  2. Consume < 2 servings of low-fat milk per day.
  3. Watch > 2 hours of TV per day.
  4. Engage in physical activity that makes them sweat or breath hard < 5 days per week.

     These behaviors have been selected because each has been associated with childhood obesity.

     5) A parent willing to attend treatment meetings. 6) Parent and child speak English.

     Exclusion Criteria:

     Participants will be excluded if they:
     1. Report a family member participating in another weight loss program.
     2. Report that the child or parent planning to attend the treatment meetings has a major psychiatric disease or organic brain syndrome.
     3. Report that the child or parent planning to attend the treatment meetings has dietary or physical activity restrictions.
     4. Intend to move outside of the metropolitan area within the time frame of the investigation.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Z-BMI in children | 12 months

SECONDARY OUTCOMES:
Eating and activity behaviors | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, Principal Investigator — University of Tennessee
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Hart CN, Raynor HA, Osterholt KM, Jelalian E, Wing RR. Eating and activity habits of overweight children on weekdays and weekends. Int J Pediatr Obes. 2011 Oct;6(5-6):467-72. doi: 10.3109/17477166.2011.590204. Epub 2011 Jul 20. PMID 21774578
- [Derived] Raynor HA, Osterholt KM, Hart CN, Jelalian E, Vivier P, Wing RR. Evaluation of active and passive recruitment methods used in randomized controlled trials targeting pediatric obesity. Int J Pediatr Obes. 2009;4(4):224-32. doi: 10.3109/17477160802596189. PMID 19922036